CLINICAL TRIAL: NCT02982928
Title: Acetaminophen Pharmacokinetics in Bariatric Patients
Brief Title: Tylenol Levels in Bariatric Patients
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Ahsan Syed, Attending Anesthesiologist, Nationwide Children's Hospital
Other Study IDs: IRB15-00471
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Obesity
Keywords: Obesity; Bariatrics; Acetaminophen; robot-assisted or laparoscopic bariatric surgery; Pharmacokinetics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The current study is designed to measure and evaluate the pharmacokinetic profiling of acetaminophen in the young obese patient population.

DETAILED DESCRIPTION:
This will be a descriptive study carried out by study staff from the anesthesiology department. The patient population will include obese patients scheduled for robot-assisted or laparoscopic bariatric surgery. There will be no change in our usual anesthetic care for these patients. Volume of distribution and elimination half-life of acetaminophen in serum samples are the primary measurements of the study. If detected, a significant reduction in opioid requirements may lead to improved patient satisfaction and decreased opiate side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 12, but younger than 21 years of age undergoing robotic assisted or laparoscopic bariatric surgery
* American Society of Anesthesiologists Physical Status Classification System (ASA) I, II or III
* Parent/guardian willing and able to give consent
* Patient willing to give assent, or consent
* Patients that are otherwise healthy at the discretion of the study staff
* Patients with BMI >95th percentile

Exclusion Criteria:

* Patients with severe right heart failure or severe asthma
* Patients with deficient hepatic function that can affect drug metabolism
* Systemic steroid use within the last 3 months
* Patients who have taken acetaminophen containing medications within 24 hours of surgery date
* Patients younger than 12, but older than 21 years of age undergoing robotic assisted or laparoscopic bariatric surgery
* Patients having other procedures in addition to robotic assisted or laparoscopic bariatric surgery
* American Society of Anesthesiologists Physical Status Classification System (ASA) IV and above
* Females testing positive for pregnancy
* Parent/guardian not willing and able to give assent, or consent
* Patient not willing to give assent, or consent
* Patients with BMI < 95th percentile

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of 30 patients presenting to the OR for robotic assisted or laparoscopic bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan Syed, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziemann-Gimmel P, Hensel P, Koppman J, Marema R. Multimodal analgesia reduces narcotic requirements and antiemetic rescue medication in laparoscopic Roux-en-Y gastric bypass surgery. Surg Obes Relat Dis. 2013 Nov-Dec;9(6):975-80. doi: 10.1016/j.soard.2013.02.003. Epub 2013 Feb 13. PMID 23499469
- [Background] Saurabh S, Smith JK, Pedersen M, Jose P, Nau P, Samuel I. Scheduled intravenous acetaminophen reduces postoperative narcotic analgesic demand and requirement after laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2015 Mar-Apr;11(2):424-30. doi: 10.1016/j.soard.2014.09.017. Epub 2014 Sep 30. PMID 25614351
- [Background] Abernethy DR, Divoll M, Greenblatt DJ, Ameer B. Obesity, sex, and acetaminophen disposition. Clin Pharmacol Ther. 1982 Jun;31(6):783-90. doi: 10.1038/clpt.1982.111. PMID 7075126
- [Background] Lee WH, Kramer WG, Granville GE. The effect of obesity on acetaminophen pharmacokinetics in man. J Clin Pharmacol. 1981 Jul;21(7):284-7. doi: 10.1002/j.1552-4604.1981.tb01768.x. PMID 7263926
- [Background] Birmingham PK, Tobin MJ, Henthorn TK, Fisher DM, Berkelhamer MC, Smith FA, Fanta KB, Cote CJ. Twenty-four-hour pharmacokinetics of rectal acetaminophen in children: an old drug with new recommendations. Anesthesiology. 1997 Aug;87(2):244-52. doi: 10.1097/00000542-199708000-00010. PMID 9286887

RESULTS

PARTICIPANT FLOW:
Groups:
- Bariatric Surgery: Obese pediatric and young adult patients undergoing robotic or laparoscopic bariatric surgery (vertical sleeve gastrectomy).
Period: Overall Study
Arm/Group | Bariatric Surgery
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bariatric Surgery
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
BMI (kg/m2) [Mean (Standard Deviation); unit: Kg/m2] | 46 (5)

OUTCOME MEASURES:

1. Primary Outcome: Intra- and Post-operative Serum Concentrations
Description: To determine whether adequate serum concentration of acetaminophen is achieved.
Time Frame: 15-20 minutes; 30-40 minutes; 50-70 minutes; 80-100 minutes; 2 Hours, 4 Hours; 8 Hours; and 12-Hours Post-IV acetaminophen administration
Measure: Mean (Standard Deviation); unit: µg.mL-1
Arm/Group | Bariatric Surgery
Number analyzed (Participants) | 11
µg.mL-1
  15-20 minutes | 17 (4)
  30-40 minutes | 14 (3)
  50-70 minutes | 9 (6)
  80-100 minutes | 5 (6)
  2 hours | 0 (0)
  4 hours | 0 (0)
  8 hours | 0 (0)
  12 hours | 0 (0)

ADVERSE EVENTS:
Time Frame: 12 hours
Arm/Group | Bariatric Surgery
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02982928/Prot_SAP_000.pdf